CLINICAL TRIAL: NCT03335410
Title: The Recuperation of Patients After Elective Shoulder Surgery -a National Observational Cohort Study
Brief Title: The Recuperation of Patients After Elective Shoulder Surgery Observational Cohort Study
Status: Completed | Type: Observational
Sponsor: Tampere University Hospital (Other)
Collaborators: Turku University Hospital (Other Government); Oulu University Hospital (Other); Kuopio University Hospital (Other); Helsinki University Central Hospital (Other); Hatanpää Hospital, Tampere (Unknown); Middle Finland Central Hospital, Jyväskylä (Unknown); Pihlajalinna, Tampere (Unknown); Terveystalo, Turku (Unknown); Satakunta Central Hospital, Pori (Unknown); Päijänne Tavastia Central Hospital (Other); Vaasa Central Hospital, Vaasa, Finland (Other)
Responsible Party: Sponsor
Other Study IDs: Kansanolka17
Record Dates: First submitted 2017-10-30; First posted 2017-11-07 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Aucte Pain After Surgery; Persistent Pain After Surgery; Opioid Use After Surgery; Mode of Anaesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- shoulder surgery: 18-85 years, undergoing day case shoulder surgery during 15th Sept- 15th Oct 2017, possibility to e-mail and an internet connection, understands Finnish,
  Interventions: Other: Non- interventional

INTERVENTIONS:
Other: Non- interventional — Non- interventional

SUMMARY:
Around 6400 shoulder surgeries are performed yearly in Finland. The procedure is mainly day-case surgery and the patients go home in the afternoon. Shoulder surgery is one of the most common procedures performed in private surgical practices. Because of the complex nature of the joint, the recovery may be complicated by severe opstoperative pain, which is relieved with strong opioids. Recently this has been addressed in the literature, as prescribed opioids too often lead to substance abuse. Pain in the acute phase after surgery is one of the common risk factors for persistent postoperative pain, which is a major burden for both the individual patient and the society.

In this prospective, observational cohort study we aim to describe current standards of practice in planning and taking care of anaeshtesia and prescribing opioids and adjuvants for postoperative pain relief at home.

DETAILED DESCRIPTION:
Around 6400 shoulder surgeries are performed yearly in Finland. The procedure is mainly day-case surgery and the patients go home in the afternoon. Shoulder surgery is one of the most common procedures performed in private surgical practices. Because of the complex nature of the joint, the recovery may be complicated by severe opstoperative pain, which is relieved with strong opioids. Recently this has been addressed in the literature, as prescribed opioids too often lead to substance abuse. Pain in the acute phase after surgery is one of the common risk factors for persistent postoperative pain, which is a major burden for both the individual patient and the society.

In this prospective, observational cohort study we aim to describe current standards of practice in planning and taking care of anaeshtesia and prescribing opioids and adjuvants for postoperative pain relief at home.

The data is collected prospectively from the care provider and the patient in a webrobol questionnaire at three time points: the day of surgery (care provider), one week after surgery (patient) and three months after surgery (patient).

ELIGIBILITY:
Inclusion Criteria:

* 18-85 years
* speaks and reads Finnish fluently
* has access to internet and email
* Undergoes elective shoulder surgery

Exclusion Criteria:

* persistent pain in an area other than the shoulder in question
* longterm pain medication for any other purpose than the shoulder in question
* schitzophrenia
* diabetes mellitus with complications

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prospective cohort of patients undergoing elective shoulder surgery and capable of answering an internet-based webropol questionnaire in Finnish.
Sampling Method: Non-Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2018-01-15 (Actual); Study Completion 2018-01-15 (Actual)

PRIMARY OUTCOMES:
Pain of the patient after shoulder surgery | 1 week after surgery
  Acute pain
wellbeing of the patient after shoulder surgery | 1 week after surgery
  well being after shoulder surgery

SECONDARY OUTCOMES:
type of anaesthesia, personnel questionnaire | Day of the surgery
  What is the anaesthesia, general anaesthesia, sedation or brachial plexus anaesthesia or a combination of these
Type of pain relief, questionnaire | 3 months after surgery
  What kind of pain relief is provided for the patients after the surgery
Persistent pain after surgery, questionnaire | three months after surgery
  How are the patients doing three months after surgery -mobility, sleep, daily habits

OTHER OUTCOMES:
Comparison of practices by a questionnaire | three months after surgery
  Compare the patient outcome results by a questionnaire based on the mode of anaesthesia/center

CONTACTS AND LOCATIONS:
Locations (14):
- Finland (14):
  - Helsinki University Hospital, Helsinki
  - Central Finland Central Hospital, Jyväskylä
  - Kuopio University Hospital, Kuopio
  - Lahti Central Hospital, Lahti
  - Oulu University Hospital, Oulu
  - Pori Central Hospital, Pori
  - Tampere University Hospital, Tampere
  - Hatanpää Hospital, Tampere
  - Pihlajalinna, Tampere
  - Pohjola Sairaala Tampere, Tampere
  - NEO Hospital, Turku
  - Terveystalo Turku, Turku
  - Turku University Hospital, Turku
  - Vaasa Central Hospital, Vaasa